CLINICAL TRIAL: NCT04750369
Title: Enhanced Triage for COVID-19 to Validate the Rapid Acute Lung Injury Diagnostic (RALI-Dx) Test
Brief Title: Enhanced Triage for COVID-19
Acronym: ETC-19
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 20-5225
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be collected in an EDTA tube for biomarker analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to evaluate of the accuracy of biomarkers (i.e. circulating endothelial and immune activation markers) that indicate progression to severe disease in patients with suspected COVID-19 in the Emergency Department. It is a prospective observational study of patients presenting to emergency departments with a clinical suspicion of COVID19. All participants will have plasma samples collected for biomarker analysis, and will be tested for SARS-CoV-2 infection with a nasopharyngeal swab. Participants will be managed according to the best local practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with clinical suspicion of COVID-19 infection, as per UHN case definition at the time of presentation
* Age >18 years
* Ability to provide verbal informed consent

Exclusion Criteria:

* Patients who are not suspected of COVID-19 infection, as per UHN definition at the time of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll patients 18 years or older, presenting to Emergency Rooms or COVID-19 Assessment Centers with clinical suspicion of COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 806 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Predictive Accuracy of Biomarkers for Risk Stratification | 28 days
  Given the expected clinical utility, we will use likelihood ratios (LRs) as our target milestone.
  +LR = (test sensitivity)/(1-test specificity);
  -LR= (1- sensitivity)/specificity.
  We will conservatively target benchmarks of +LR>5 for a disposition towards and a -LR<0.1 for a disposition away from mortality risk.

SECONDARY OUTCOMES:
Performance of Biomarkers as Indicators of Clinical Severity: Disposition post-ED visit (admitted vs discharged home vs discharged home and readmitted) | 28 days
Performance of Biomarkers as Indicators of Clinical Severity: Hospital and ICU length of stay | 28 days
Performance of Biomarkers as Indicators of Clinical Severity: Need for artificial respiratory support or hemodynamic support (mechanical ventilation, ECLS) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Husain, MD MS, Principal Investigator — University Health Network, Toronto
Locations (3):
- Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Brazil
- University Health Network, Toronto, Ontario, Canada
- Cittá della Salute e della Scienza di Torino Hospital-Molinette Site, Turin, Italy

IPD SHARING:
Plan to Share IPD: No